CLINICAL TRIAL: NCT02980159
Title: Impact of a Triage Liaison Physician on the Time to First Medical Evaluation in the Emergency Departement
Brief Title: Impact of a Triage Liaison Physician
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Olivier T. Rutschmann, Professor, Chief deputy, University Hospital, Geneva
Other Study IDs: CCER 2016-00179
Record Dates: First submitted 2016-11-24; First posted 2016-12-02 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Emergencies; Triage
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Before triage liaison physician: All patients admitted before the introduction of the function of triage liaison physician.
- After triage liaison physician: All patients admitted after the introduction of the function of triage liaison physician.
  Interventions: Other: Triage liaison physician

INTERVENTIONS:
Other: Triage liaison physician — A triage liaison physician is present from 7:30 am to 10:30 pm, Monday to Friday, with the mission to evaluate quickly patients who cannot be immediately installed in an ED room
  Groups: After triage liaison physician

SUMMARY:
Due to an increasing number of patients admitted in emergency departments, many patients cannot be evaluated immediately after their admission. The function of "triage liaison physician" was introduced in Spring 2015. The objective of this study is to evaluate the impact of this new function on patients' flow in the ED.

DETAILED DESCRIPTION:
Geneva University Hospitals (GUH) emergency department (ED) admits more than 64000 patients every year. These patients are triaged using the Swiss Emergency Triage Scale (SETS), a 4-level triage scale. The SETS imposes time objectives until the first medical evaluation (20 minutes for SETS 2, 2 hours for SETS 3). In 2014, only 60% of level-2 and 63% of level-3 emergencies were evaluated within 20 and 120 minutes respectively.

A triage liaison physician was introduced in Spring 2015 with the mission to help triage nurse in their decisions and to evaluate quickly the patients that cannot be immediately installed in an ED evaluation room.

The objective of this study is to evaluate the impact of the triage liaison physician on the times to first medical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* >= 16 y
* admitted in GUH ED

Exclusion Criteria:

* patients triaged to outpatient clinics

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patient admitted in GUH ED during 2 years.
Sampling Method: Non-Probability Sample
Enrollment: 69893 (Actual)
Dates: Start 2016-11; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients evaluated within SETS objectives | Within 120 minutes after ED triage
  Proportion of patients evaluated within time objective as defined by SETS standards.

SECONDARY OUTCOMES:
Time to first medical contact | Within 24 hours after ED triage
  Time elapsed between triage and first medical evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Olivier T Rutschmann, MD, MPH, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals, ED, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No